CLINICAL TRIAL: NCT05480592
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Phase I Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of HS-10380 in Chinese Healthy Adult Subjects
Brief Title: A Study of HS-10380 in Chinese Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-10380-101
Record Dates: First submitted 2022-07-05; First posted 2022-07-29 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; HS-10380
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (SAD) (Experimental): Subjects in cohorts 1-6 will receive oral administration of single dose of HS-10380 tablets or matching placebo.
  Interventions: Drug: HS-10380; Drug: Placebo
- Multiple Ascending Dose (MAD) (Placebo Comparator): Subjects in cohorts 7 will receive oral administration of 7 dose of HS-10380 tablets or matching placebo.
  Interventions: Drug: HS-10380; Drug: Placebo

INTERVENTIONS:
Drug: HS-10380 — Administered orally as a tablet
Drug: Placebo — Administered orally as a tablet

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of single and multiple oral administered doses of HS-10380 in Chinese healthy subjects.

DETAILED DESCRIPTION:
This is a phase I, randomized, double-blinded, placebo-controlled, both single ascending doses (SAD) study and multiple ascending dose (MAD) clinical trial to assess the safety, tolerability, and pharmacokinetics of HS-10380 in Chinese healthy subjects.

There will be four phases in SAD and MAD study: a 2-week screening phase, a 1-day baseline phase, a double-blind treatment phase, and a 1-week post-treatment (follow-up) phase.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject aged from 18 to 45 years;
2. Subject has a Body Mass Index (BMI) between 18.5 and 26.0 kg/m2 at screening and the weight of male subjects is not less than 50 kg, and the weight of female subjects is not less than 45 kg;
3. Voluntary subject who signs the informed consent form after understanding the purpose, content, process and possible risks of the trial;
4. Subject is able to communicate well with the investigator and comply with the lifestyle constraints specified in the protocol, and cooperate to complete the trial procedures.

Exclusion Criteria:

1. Subject has history or presence of disease or dysfunction affecting the clinical trial, including but not limited to neuropsychiatric system, cardiovascular system, urinary system, digestive system, respiratory system, musculoskeletal system, metabolic endocrine system, skin disease, blood system disease, immune system and tumor, etc.;
2. Subject has any surgical condition or condition that may significantly affect the absorption, distribution, metabolism, and excretion of the drug, or any surgical condition or condition that may pose a hazard to the subjects participating in the trial, such as gastrointestinal surgery (gastrectomy, Gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or dysuria, gastroenteritis, peptic ulcer, history of gastrointestinal bleeding, etc.;
3. Subject has a history of significant drug allergies or known allergies to the components of the test drug;
4. Subject has history or presence of psychiatric disorders and cerebral dysfunction, or subjects at risk of suicide according to the Columbia Suicide Severity Rating Scale (C-SSRS) or at risk of suicide according to the investigator's clinical judgment, or has a history of self-harm;
5. Subject has a history of drug abuse within 1 year prior to screening, or has a positive urine drug result screen at screening;
6. Subject has history of alcohol abuse or a single consumption of more than 14 units of alcohol (1 unit = 285 mL of beer, 25 mL of spirits, 150 mL of wine) in the nearly one year prior to screening or a positive breath test for alcohol at screening;
7. Subject has smoked ≥5 cigarettes per day or consumed an average of ≥5 (200mL/cup) cups of coffee or tea per day in the 3 months before screening, or could not stop users during the study;
8. Subject has special requirements for food or is unwilling to accept a uniform diet or has difficulty swallowing;
9. Pregnant or breastfeeding women, or those who refuse to use effective contraception (eg, abstinence, IUD) throughout the study period and 6 months after the end of the study, or those who have a sperm or egg donation plan;
10. Subject has clinically significant abnormal comprehensive physical examination, vital signs, laboratory tests, and 12-lead electrocardiograms, which are judged by the investigator (eg: QTcF>450ms for men and >470ms for women, Friericia correction);
11. Subject with resting pulse rate <55 bpm or >100 bpm; systolic blood pressure <90mmHg or >140mmHg; diastolic blood pressure <60mmHg or >90mmHg at screening;
12. Subject has detectable hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV), or human immunodeficiency virus (HIV) antibody at screening;
13. Subject with alanine aminotransferase (ALT), creatinine (Cr), blood urea nitrogen (BUN) exceeding the upper limit of normal or serum prolactin greater than 2 times the upper limit of normal at the time of screening;
14. Subject has donated blood or lost blood ≥ 400ml within 3 months before screening, or donated blood or lost blood ≥ 200ml within one month, or has a history of using blood products;
15. Subject with a history of surgery within 3 months prior to screening, or who have not recovered from surgery, or who have anticipated surgery plans during the trial;
16. Subject has taken any medication within 2 weeks (or 5 half-lives, whichever is longer) prior to screening or takes any medication throughout study, including prescription and over-the-counter medications, Chinese herbal medicines, and any drugs that inhibit or induce liver drug metabolizing enzymes (such as inducers and/or inhibitors of CYP3A4, CYP2D6 and CYP3A5);
17. Subject has participated in any clinical trial or took any clinical trial drugs within 3 months before screening;
18. Subject has dieted or received dietary therapy, or had significant changes in dietary habits within 30 days prior to screening;
19. Subject has a history of vaccination within 30 days prior to screening, or has a vaccination schedule throughout the study;
20. Subject with poor compliance or other problems which the investigator considers unsuitable for subject to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects Experiencing Adverse Events (AEs) | Baseline to end of follow-up (a maximum of 20 days)
  AE include adverse events (AEs) and serious adverse events (SAEs)
Changes from baseline in laboratory tests | Baseline to end of follow-up (a maximum of 20 days)
  Laboratory tests include blood routine, urine routine, blood biochemistry, coagulation function, thyroid function and serum prolactin;
Changes from baseline in vital signs | Baseline to end of follow-up (a maximum of 20 days)
  Vital signs include respiration, pulse, blood pressure, body temperature and SpO2
Change from baseline in Electrocardiogram (ECG) | Baseline to end of follow-up (a maximum of 20 days)
  ECG parameters including heart rate, PR interval, RR interval and QTcF, etc.
Change from baseline in weight (kg) | Baseline to end of follow-up (a maximum of 20 days)
Change from baseline in physical examination | Baseline to end of follow-up (a maximum of 20 days)
  Including general condition, heart, chest and abdomen, skin and mucous membranes, lymph node examination, etc.
Change from baseline in Simpson-Angus Scale (SAS) score | Baseline to end of follow-up (a maximum of 20 days)
  The SAS is a 10-item testing instrument used to evaluate drug-related extrapyramidal syndromes. The following items are included in the SAS: gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head dropping, glabella reflex, tremor, and salivation. Total score ranges from 0 to 40 with a higher score indicating increased severity.
Change from baseline in Abnormal Involuntary Movement Scale (AIMS) score | Baseline to end of follow-up (a maximum of 20 days)
  AIMS is a rating scale measuring involuntary movements known as tardive dyskinesia, that sometimes develop as a side effect of long-term treatment with antipsychotic medications. The AIMS score was calculated as the sum of questions 1 through 7 of the AIMS instrument, which includes assessments of involuntary movements in the face, lips, jaw, tongue, upper and lower extremities, and neck/shoulders/hips. Each item is rated on a five-point scale of severity from 0-4 with 0 (none), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe). Total scores range from 0 to 28.
Change from baseline in Barnes Akathisia Rating Scale (BARS) score | Baseline to end of follow-up (a maximum of 20 days)
  BAS is a rating scale that is administered by physicians to assess the severity of drug-induced akathisia, which is a movement disorder characterized by a feeling of inner restlessness and a compelling need to be in constant motion, as well as by actions such as rocking while standing or sitting, lifting the feet as if marching on the spot, and crossing and uncrossing the legs while sitting. The following subcategories are scored: objective akathisia, subjective awareness of restlessness and subjective distress related to restlessness and are rated on a 4-point scale from 0-3. In addition, the global clinical assessment of akathisia uses a 6-point scale ranging from 0-5. Total score ranges from 0 to 14 with a higher score indicating increased severity.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of single-dose HS-10380 administration | Up to 120 hours post-dose
Time of the Maximum Concentration (Tmax) of single-dose HS-10380 administration | Up to 120 hours post-dose
Terminal rate constant (λz) of single-dose HS-10380 administration | Up to 120 hours post-dose
Elimination half-life (t1/2) of single-dose HS-10380 administration | Up to 120 hours post-dose
Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC0-t) of single-dose HS-10380 administration | Up to 120 hours post-dose
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC0-∞) of single-dose HS-10380 administration | Up to 120 hours post-dose
Apparent clearance (CL/F) of single-dose HS-10380 administration | Up to 120 hours post-dose
Apparent volume of distribution (Vd/F) of single-dose HS-10380 administration | Up to 120 hours post-dose
Mean retention time (MRT) of single-dose HS-10380 administration | Up to 120 hours post-dose
Maximum plasma concentration (Cmax) of first HS-10380 administration | Up to 12 days
Time of the Maximum Concentration (Tmax) of first HS-10380 administration | Up to 12 days
Area under the plasma concentration-time curve from time zero to 24 hours (AUC0-24) first HS-10380 administration | Up to 24 hours
Maximum concentration at steady state (Css, max) of multiple-dose HS-10380 administration | Up to 12 days
Time of the maximum concentration at steady state (Tss, max) of multiple-dose HS-10380 administration | Up to 12 days
Minimum concentration at steady state (Css, min) of multiple-dose HS-10380 administration | Up to 12 days
Area under the concentration-time curve at steady state (AUCss) of multiple-dose HS-10380 administration | Up to 12 days
Accumulation ratio (RAC) after multiple doses | Up to 12 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China